CLINICAL TRIAL: NCT00017654
Title: Study of Allogeneic Bone Marrow and T-Cell Depleted, CD34+ Peripheral Blood Stem Cell Transplantation in Patients With Aplastic Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern Memorial Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14983; NU-96AA1T; NU-96H
Record Dates: First submitted 2001-06-06; First posted 2001-06-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Graft Versus Host Disease; Aplastic Anemia
Keywords: aplastic anemia; disease-related problem/condition; graft versus host disease; hematologic disorders; rare disease
MeSH Terms: conditions — Graft vs Host Disease; Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; Methylprednisolone

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methylprednisolone
Procedure: Allogeneic Bone Marrow Transplantation

SUMMARY:
OBJECTIVES:

I. Determine the effect of supplementation with donor T-cell depleted, CD34+ peripheral blood stem cells on durable engraftment and incidence of graft-versus-host disease in patients with aplastic anemia undergoing allogeneic bone marrow transplantation.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Bone marrow and peripheral blood stem cells (PBSC) are harvested from a HLA identical or 1 antigen mismatched related donor. PBSC are selected for CD34+ cells and T cells are depleted.

Patients receive cyclophosphamide IV over 2 hours on days -6 to -3 and anti-thymocyte globulin IV with methylprednisolone IV over 10-12 hours on days -5 to -3. T-cell depleted PBSC and bone marrow are infused on day 0. Patients receive cyclosporine IV over 12-24 hours on days -1 to 120 followed by a taper and methylprednisolone IV on days 7-64 for graft-versus-host disease prophylaxis.

Patients are followed every 30 days for 1 year, every 60 days for 2 years, and then as needed for a minimum of 3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of life-threatening or transfusion-dependent marrow or immune-mediated failure involving one or more hematopoietic cell lines evidenced by one or more of the following: Granulocyte count less than 500/mm3 Platelet count less than 20,000/mm3 Absolute reticulocyte count less than 60,000/mm3
* Immune-mediated anemia and/or thrombocytopenia must have failed corticosteroids and cyclosporine
* Paroxysmal nocturnal hemoglobinuria with progressive marrow failure allowed
* Either congenital or acquired severe granulocytopenia with a history of life threatening infections No diagnosis of Fanconi's anemia
* HLA identical or 1 antigen mismatched related donor meeting the following criteria: No prior or concurrent malignancy except localized basal cell or squamous cell skin cancer (malignancies judged to be cured by local surgery, such as head and neck cancer or stage I breast cancer, considered on an individual basis) Negative pregnancy test

--Patient Characteristics--

* Hepatic: Hepatitis B surface antigen negative Bilirubin no greater than 2.0 mg/dL Transaminases no greater than 2 times upper limit of normal (in the absence of Gilbert's disease)
* Renal: Creatinine no greater than 2.0 mg/dL
* Cardiovascular: No history of coronary artery disease LVEF at least 40% by MUGA
* Pulmonary: FEV1 at least 50% predicted FVC at least 50% predicted DLCO at least 50% predicted
* Other: No uncontrolled diabetes mellitus No other illness that would preclude aggressive chemotherapy No prior or concurrent malignancy except localized basal cell or squamous cell skin cancer (malignancies judged to be cured by local surgery, such as head and neck cancer or stage I breast cancer, considered on an individual basis) No psychiatric illness or mental deficiency that would preclude study Not pregnant or nursing Fertile patients must use effective contraception HIV negative

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Burt, Study Chair — Northwestern Memorial Hospital
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States